CLINICAL TRIAL: NCT02796196
Title: Effects of Prescribed Physical Activity on Sleep and Performance in Hematopoietic Cell Transplantation Patients
Brief Title: Prescribed Physical Activity in Improving Sleep and Physical Performance in Patients Undergoing Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-35379; NCI-2016-00737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VAR0137 (Other: Stanford Cancer Institute); IRB-35379 (Other: Stanford IRB)
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Cell Transplantation
Keywords: Hematopoietic; Recipient
MeSH Terms: interventions — Monitoring, Physiologic; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive care (monitoring device, medical chart review): Data including demographics, type of HCT (e.g., allogeneic or autologous), preexisting physical conditions (e.g., chronic joint injury), CRF, steroid use data, ECOG and KPS scores are collected from patients' medical charts at time of enrollment. Patients are prescribed participation in a primarily self-directed physical activity program which encourages them to spend 6 hours out of bed daily and to perform 30 minutes of light-to-moderate daily aerobic activity. Patients who are able to maintain independent mobility undergo physical therapist assessment 2 times a week until hospital discharge. Patients wear a physical activity monitoring device and daily activity and sleep data are collected continuously during hospital LOS.
  Interventions: Other: Medical Chart Review; Device: Monitoring Device; Procedure: Physical Therapy

INTERVENTIONS:
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Device: Monitoring Device — Wearable physical activity monitoring device
  Other Names: Monitor
Procedure: Physical Therapy — Undergo primarily self-directed physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT

SUMMARY:
This research trial studies prescribed physical activity in improving sleep and physical performance in patients undergoing stem cell transplant. A wearable physical activity monitor can be used to record minutes of activity and sleep. Gathering data over time using a physical activity monitor may help doctors learn if prescribed physical activity helps improve sleep and physical performance in patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate whether prescribed physical activity, as part of standard care, improves sleep and functional outcomes in hematopoietic cell transplantation (HCT) (stem cell transplantation) patients during a typical 30-day hospitalization period.

OUTLINE:

Data including demographics, type of HCT (e.g., allogeneic or autologous), preexisting physical conditions (e.g., chronic joint injury), chronic renal failure (CRF), steroid use data, Eastern Cooperative Oncology Group (ECOG) and Karnofsky performance status (KPS) scores are collected from patients' medical charts at time of enrollment. Patients are prescribed participation in a primarily self-directed physical activity program which encourages them to spend 6 hours out of bed daily and to perform 30 minutes of light-to-moderate daily aerobic activity. Patients who are able to maintain independent mobility undergo physical therapist assessment 2 times a week until hospital discharge. Patients wear a physical activity monitoring device and daily activity and sleep data are collected continuously during hospital length of stay (LOS).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Stanford Hospital for HCT
* Able to provide informed consent
* Speaks language supported by interpretative services
* Able to operate and take care of a physical activity monitor

Exclusion Criteria:

* Does not meet inclusion criteria
* Unable to wear a physical activity monitor throughout hospital stay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Stem Cell Transplant at Stanford Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
ECOG performance scores | At baseline
  Will focus on trends in scores between patients with different durations of activity and sleep. Results, from both descriptive and inferential analyses, will be presented in table and/or graphical format.
KPS performance scores | At baseline
  Will focus on trends in scores between patients with different durations of activity and sleep. Results, from both descriptive and inferential analyses, will be presented in table and/or graphical format.
Minutes of aerobic activity per day | Up to time of hospital discharge, or 29 days
  Will use interval-censored regression to estimate distributions of activity from one day to the next. This repeated-measures analysis with a polynomial model will generate average curves for activity, each spanning average LOS (i.e., activity duration plotted on day one, day two, day three, etc.). Will also run diagnostics to verify the assumptions of a linear model (e.g., statistical independence of observations and lack of undue influence of outliers on model fit).
Minutes of sleep per day | Up to time of hospital discharge, or 29 days
  Will use interval-censored regression to estimate distributions of sleep from one day to the next. This repeated-measures analysis with a polynomial model will generate average curves for sleep, each spanning average LOS (i.e., sleep duration plotted on day one, day two, day three, etc.). Will use multiple linear regressions to control for potential confounders in predicting sleep duration. Will also run diagnostics to verify the assumptions of a linear model (e.g., statistical independence of observations and lack of undue influence of outliers on model fit).

CONTACTS AND LOCATIONS:
Overall Officials: André Valdez, Principal Investigator — Stanford University; Matthew Smuck, Principal Investigator — Stanford University; Kota Reichert, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No